CLINICAL TRIAL: NCT00113464
Title: Developing Newborn Screening for Infants With Primary Immunodeficiency
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050162; 05-HG-0162
Record Dates: First submitted 2005-06-07; First posted 2005-06-08 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-04-13

CONDITIONS: Immune System Diseases
Keywords: SCID (Severe Combined Immunodeficiency); TREC (T cell Receptor Excision Circle); Bone Marrow Transplant; Dried Blood Spots; Early Detection; T Cell Immunodeficiency Diseases; Immunodeficiency Diseases; Primary Immunodeficiency; T Cell Immunodeficiency Disease; Severe Combined Immunodeficiency; SCID
MeSH Terms: conditions — Immune System Diseases; X-Linked Combined Immunodeficiency Diseases; Primary Immunodeficiency Diseases; Severe Combined Immunodeficiency

SUMMARY:
This study will explore screening for immunodeficiency diseases (diseases that cause problems in fighting infections). There is no method at present to screen all babies at birth for immunodeficiency. However, babies with low numbers of T-cells-an important type of immune system cell-may be found by studying T-cell products called TRECs (T-cell receptor excision circles). This study will:

* Collect samples from children with several different immunodeficiencies to find out which disorders can be found by screening dried blood spots for TRECs.
* Try to develop screening tests based on other kinds of material derived from dried blood spots.

Children with primary immunodeficiency and low numbers of T cells who have not had a bone marrow transplant may be eligible for this study.

Participating children donate up to 5 ml (1 teaspoon) of blood. The sample may be collected when the child is having other blood tests. The liquid blood is analyzed to determine the number of T cells, and the rest of the blood is used to make dried blood spots on filter paper. The blood spots are used to develop screening tests for immunodeficiency. The blood spots and data about the child's age, diagnosis, and current medicines will be kept coded by diagnosis and a code number instead of the child's name.

DETAILED DESCRIPTION:
Study Objective: T cell receptor excision circles (TRECs) are episomal DNA circles excised from the T cell receptor genes during T cell maturation in the thymus. They do not replicate, so they are diluted out as T cells proliferate. Our objectives are to examine the levels of TRECs in blood samples from patients with primary immunodeficiency (PI) diseases; to determine which PI diseases might be detected by testing newborn dried blood spots for low numbers of TRECs; and to use the blood spots collected for future confirmatory or alternative tests to develop newborn screening for PIs.

Population: Patients diagnosed with defined primary T cell immunodeficiency diseases or undefined conditions with very low T cell numbers. There are several known, and additional unknown, gene defects that impair T lymphocyte maturation and function. The frequency of these rare disorders is unknown, but could potentially be learned in the course of population-based newborn screening.

Design: We will contact our network of immunology colleagues to help us identify and enroll patients already diagnosed with PI disorders. These patients will have had HIV ruled out as part of their immune evaluation. We will provide mail-in kits and will receive blood samples for analysis. We will attempt to retrieve the actual Guthrie cards containing the dried blood spots of these patients from their state screening laboratories to determine the number of TRECs that were present at birth in infants with these conditions.

Outcome Measures: We will measure TRECs in dried blood spots, and correlate TREC number with diagnosis and clinical and laboratory data. We hope to determine the range of immunodeficiency diseases that can be demonstrated to have significantly reduced TRECs as compared to healthy subjects using our assay. Because TREC testing may be insufficiently sensitive or specific as a stand-alone test, further tests may be developed and performed on the samples in the future, including DNA re-sequencing, detection of mRNA for T cell specific genes and/or proteins expressed only in T cells.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patient who has not yet received a BMT and who has defined PI or undefined PI with T cell lymphopenia.

EXCLUSION CRITERIA:

None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2005-06-02; Study Completion 2007-04-13

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Background] Barrett DJ, Ammann AJ, Wara DW, Cowan MJ, Fisher TJ, Stiehm ER. Clinical and immunologic spectrum of the DiGeorge syndrome. J Clin Lab Immunol. 1981 Jul;6(1):1-6. PMID 6973633